CLINICAL TRIAL: NCT03808246
Title: Detection of Usability Errors of a Medical Device Zeneo®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017_16; 2017-A02847-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-09-18; First posted 2019-01-17 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: 2 profiles of participants (naïves vs. informed) x 2 types of test environment (realistic vs. laboratory-like).
  Each participant, depending on her/his profile is assigned to one "profile of participant" group and randomly to one "type of test environment" group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- naive/realistic environment (Experimental): This arm includes included participants who are naive in terms of self-injector pens and who have been randomly attributed to the "realistic environment" condition of simulation.
  The intervention is "using the demo version of a self-injector pen".
  Interventions: Other: using the demo version of a self-injector pen
- informed/realistic environment (Experimental): This arm includes included participants who are informed in terms of self-injector pens and who have been randomly attributed to the "realistic environment" condition of simulation.
  The intervention is "using the demo version of a self-injector pen".
  Interventions: Other: using the demo version of a self-injector pen
- informed/laboratory-like environment (Experimental): This arm includes included participants who are informed in terms of self-injector pens and who have been randomly attributed to the "laboratory-like environment" condition of simulation.
  The intervention is "using the demo version of a self-injector pen".
  Interventions: Other: using the demo version of a self-injector pen
- naive/laboratory-like environment (Experimental): This arm includes included participants who are naive in terms of self-injector pens and who have been randomly attributed to the "laboratory-like environment" condition of simulation.
  The intervention is "using the demo version of a self-injector pen".
  Interventions: Other: using the demo version of a self-injector pen

INTERVENTIONS:
Other: using the demo version of a self-injector pen — Participants, whatever the arm they are included in, will have to use the demo version of the auto-injector pen during a simulation of an anaphylactic shock.

SUMMARY:
The research addresses the question of the number of participants needed to identify as many usability-induced errors as possible in the context of summative usability tests. The research addresses also the impact of the ecological validity of the test environment on the number of usability-induced errors uncovered.

DETAILED DESCRIPTION:
In order to determine how many participants must be recruited to detect 95% of the anticipated use errors, two groups of participants (naives or informed to the type of device under evaluation) will take part to usability test of a demo version of an auto injector pen in one of two test environments (realistic or laboratory-like). The combination of the 2 types of users and the two types of environment composes 4 arms.

By default, 15 participants will be recruited per arm (in conformity with usual guidelines). If, in a given group, 95% of anticipated errors are detected, no more participants will be recruited in the arm. Otherwise, 5 other participants will be recruited till the 95% threshold is reached with a maximum of 40 participants per group.

ELIGIBILITY:
Two types of participants (healthy people) will be recruited: participants informed about auto-injector pens (BUT NOT PATIENTS) and participants naïves on this topic.

Inclusion Criteria:

* Able to use the device
* Without previous experience of anaphylactic shock
* Not taking a psychotropic drug
* Without hearing impairment
* Covered by social security
* Who signed the consent form and the information letter
* Who agree to conform to the procedure of the study -

Exclusion Criteria:

* Pregnant women
* Vulnerable Persons
* Persons under administrative supervision
* Persons who are subject to a judicial protection measure
* Persons who do not understand correctly French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
For each arm, number of participants needed to uncover 95% of the use errors known | through study completion, an average of 6 months

SECONDARY OUTCOMES:
number of use errors uncovered per participant | through study completion, an average of 6 months
number of participants who detected a given error | through study completion, an average of 6 months
number of unanticipated errors detected | through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Romaric Marcilly, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Usability Lab of CIC IT 1403, Lille, Haut de France, France